CLINICAL TRIAL: NCT06728345
Title: The Real-world Study of Rimegepant for the Preventive Treatment in Female Migraine Patients
Brief Title: The Real-world Study of Rimegepant Treatment in Female Migraine Patients of China
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: No.2024-454
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Migraine; Migraine Prophylaxis
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- female migraine patients who recevie Rimegepant as prophylactic treatment
  Interventions: Drug: Rimegepant

INTERVENTIONS:
Drug: Rimegepant — Female migraine patients take Rimegepant (75mg QOD) as their regular prophylactic treatment of migraine for 12 weeks

SUMMARY:
The goal of this observational study is to learn about the effects and safety of Rimegepant in women, especially young and middle-aged women, who take Rimegepant to treat their migraine in the real world. Participants already taking Rimegepant (75mg QOD) as their regular preventive treatment of migraine for 12 weeks will be evaluated as the followings :

1. To evaluate the change from baseline in the mean number of migraine days per month during weeks 1-12
2. To evaluate the number of participants that have least a 50% reduction from baseline in the mean number of migraine days per month during weeks 1-12

DETAILED DESCRIPTION:
This single arm, prospective, multi-center, observational registry study aim to evaluate effectiveness of rimegepant as preventive migraine treatment in the real-world setting.

About 300 adult migraine participants will be enrolled continuously at 6 sites with a headache clinic or headache center in China. Subjects who meet the inclusion criteria will be enrolled and will participate in the study. Baseline data including demographic information, socio-economic information, physical examination, medical history, migraine history and past use of headache medications will be collected at the baseline visit. The treatment period will last for 12 weeks during which patients will take rimegepant 75 mg orally disintegrating tablet every other day. The efficacy of rimegepant measured by the reduction in the number of migraine days per month. Subjects will be asked to keep a headache diary to collect monthly headache and migraine days, migraine severity, associated symptoms and drug consumption. Data will be collected at baseline and every month. At study visits, participants will complete the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder -7 (GAD-7), Headache Impact Test-6 (HIT-6), Pittsburgh Sleep Quality Index (PSQI) at weeks 4, 8 and 12; and participants will complete the Migraine Disability Assessment (MIDAS) at weeks 12.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants aged ≥ 18 years-old
2. Primary diagnosis of migraine according to ICHD-3 3.4 or more migraine days during Observation Period and Screening Visit

4.Migraine attacks present for more than 1 year 5.Rimegepant is prescribed for the preventive treatment of migraine by physician 6.Written informed consent must be obtained before participant is enrolled 7.Not concurrently participating in other interventional clinical studies.

Exclusion Criteria:

1. Patients diagnosed with secondary headaches.
2. Women who are pregnant or breastfeeding.
3. Subjects with severe impairments in language, vision, memory, or cognitive function that affect communication and understanding, or those who are unable to complete questionnaires or follow-ups.
4. Subjects lacking the equipment to complete questionnaires on a digital platform.
5. Subjects who are allergic to rimegepant or any of its excipients.
6. Patients with severe liver damage or end-stage renal disease.
7. Patients with a medical history indicating the presence of uncontrolled or unstable cardiovascular disease (such as ischemic heart disease, coronary artery spasm, or cerebral ischemia), or those who have had a myocardial infarction, acute coronary syndrome, percutaneous coronary intervention, cardiac surgery, stroke, or transient ischemic attack within 6 months prior to the screening visit.
8. Any condition deemed by the investigator that might affect the patient's participation in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients diagnosed with migraine (with or without aura) who take rimegepant rimegepant 75 mg orally disintegrating tablet every other day for 12 weeks
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from the baseline in the number of migraine days per month over the entire treatment phase (Weeks 1-12) | The treatment period is 12 weeks
  Change from baseline in mean number of migraine days per month
Proportion of subjects with > 50% reduction from the baseline (Weeks 1 to 12) | The treatment period is 12 weeks
  Number of migraine days per month over the entire treatment phase

SECONDARY OUTCOMES:
Mean change from the baseline in the number of moderate or severe migraine days per month over the entire treatment phase (Weeks 1-12) | The treatment period is 12 weeks
  Change from baseline in mean number of moderate or severe migraine days per month
Mean change from baseline in the Migraine Disability Assessment (MIDAS) | Baseline, Week 12
  Changes in MIDAS score across rimegepant treatment. Participants provide the number of missed work or school days; missed household chores days; missed social or leisure activity days; and days at work or school, and separately at home, where productivity was reduced by half or more in the last 3 months (scale: 0 - 90 for each of 5 subscales). The 5 subscale scores are summed to compute the MIDAS total score (scale: 0 - 450). Lower scores indicate less headache-related disability.
Mean change from baseline in the migraine disability (HIT-6) | Baseline , Week 4,8,12
  Changes in Headache Impact Test-6 questionnaire across rimegepant treatment. Headache Impact Test (HIT-6) is a measure of headache severity and provides information regarding the effect of headache on other domains related to functional participation. The HIT-6 has six questions and the range goes from 36 (best outcome) to a maximum score of 78 (worst outcome). Higher HIT-6 scores indicate increased headache severity and greater functional limitations
Mean change from baseline in the Patient Health Questionnaire (PHQ-9) | Baseline , Week 4,8,12
  Changes in PHQ-9 questionnaire across rimegepant treatment. PHQ-9 scoring uses a 4-point Likert scale: 0 = "Not at all," 1 = "Some days," 2 = "More than half the days," and 3 = "Almost every day." With a total score ranging from 0 to 27
Mean change from baseline in the Generalized Anxiety Disorder -7 (GAD-7) | Baseline , Week 4,8,12
  Anxiety level is measured with Generalized Anxiety Disorder 7-item (GAD-7) which is a tool based on seven items which are scored from zero to three. The whole scale score can range from 0 to 21 and cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively
Mean change from baseline in the Pittsburgh Sleep Quality Index (PSQI) | Baseline , Week 4,8,12
  Changes in PSQI questionnaire across rimegepant treatment. PSQI is a self-rated questionnaire for sleep quality. It includes 18 items across 7 components; C1: Sleep quality, C2: Sleep latency, C3: Sleep duration, C4: Sleep efficiency, C5: Sleep

IPD SHARING:
Plan to Share IPD: No